CLINICAL TRIAL: NCT01581476
Title: Randomised, Double Blind, Placebo Controlled Trial of Angiotensin Converting Enzyme Inhibitors and Statins in the Prevention of Long Term Complications in Young People With Type 1 Diabetes
Brief Title: Adolescent Type 1 Diabetes Cardio-Renal Intervention Trial
Acronym: AdDIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Diabetes UK (Other); British Heart Foundation (Other); Pfizer (Industry); The University of Western Australia (Other); The Hospital for Sick Children (Other); University of Oxford (Other); St Thomas' Hospital, London (Other)
Responsible Party: Principal Investigator, David Dunger, Professor David Dunger, University of Cambridge
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: RP06; 2007-001039-72 (EudraCT Number)
Record Dates: First submitted 2012-04-13; First posted 2012-04-20 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes
Keywords: Adolescence
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Angiotensin-Converting Enzyme Inhibitors; Quinapril; Combined Modality Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Statin (Active Comparator): Participants receive active statin and placebo ACE Inhibitor
  Interventions: Drug: Statin
- Angiotensin-converting enzyme inhibitor (Active Comparator): Participants receive active ACE Inhibitor and placebo statin
  Interventions: Drug: ACE inhibitor
- Placebo (Placebo Comparator): Participants receive placebo ACE Inhibitor and placebo statin
  Interventions: Drug: Placebo
- Combination therapy (Other): Participants receive both active ACE Inhibitor and active Statin
  Interventions: Drug: Combination therapy

INTERVENTIONS:
Drug: Statin — 10mg daily for a minimum period of 2 years
  Other Names: Atorvastatin
  Arms: Statin
Drug: ACE inhibitor — Starting dose of 5mg daily rising after 14 days to 10mg daily providing it is well tolerated for a minimum period of 2 years.
  Other Names: Quinapril
  Arms: Angiotensin-converting enzyme inhibitor
Drug: Placebo — Participants receive statin placebo and ACEI placebo
  Arms: Placebo
Drug: Combination therapy — Participants receive both active statin and active ACEI. Dose for Statins is 10mg daily. Dosing for ACEI starts at 5mg daily rising to 10mg after 14 days providing it is well tolerated. Both interventions last for a minimum of 2 years.
  Other Names: Atorvastatin; Quinapril
  Arms: Combination therapy

SUMMARY:
The purpose of this study is to determine whether use of blood pressure lowering drugs, Angiotensin converting enzyme inhibitors (ACEIs) and blood fat (lipid) lowering drugs (statins) may have a place in the treatment of adolescents with diabetes and can help reduce serious long-term health problems in this population.

DETAILED DESCRIPTION:
Subjects will be recruited from a pre-screened population of 3,000 young people with T1D aged 10 to 16 years based on assessment of risk for future CVD and DN.

They will be randomised to a 2 x 2 factorial design contrasting the effects of ACEI, statins, or combination therapy to placebo over a maximum four year treatment period. Minimisation of variation in albumin excretion rate, gender, age, diabetes duration, HbA1c, total cholesterol and centre site will be undertaken at randomisation.

Analysis of the primary endpoint, change in albumin excretion will be undertaken on an intention to treat basis. Secondary analyses will be undertaken on the basis of 'as treated' allowing for variance in compliance and allowing for subjects who show substantial change in HbA1c levels. Additional analyses will be undertaken to assess changes in the secondary objectives and to assess the overall effect of the intervention on quality of life and health economics.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10 to 16 years.
2. T1D diagnosed for more than 1 year or C-peptide negative.
3. Centralised assessment of ACR based on six early morning urines deemed to be in upper tertile for risk after adjustment for age, gender, age at diagnosis and duration of disease.

Exclusion Criteria:

1. Non T1D, i.e. type 2 diabetes, insulin dependent diabetes related to monogenic disease, secondary diabetes.
2. ACR based on six early morning urines deemed to be at low risk for subsequent development of CVD or DN.
3. Pregnancy or unwillingness to comply with contraceptive advice and regular pregnancy testing throughout the trial.
4. Breast feeding
5. Severe hyperlipidaemia and family history data to support diagnosis of familial hypercholesterolaemia.
6. Established hypertension unrelated to DN.
7. Prior exposure to the investigational products, statins and ACEI.
8. Unwillingness/inability to comply with the study protocol.
9. Other co-morbidities considered unsuitable by the investigator (excluding treated hypothyroidism and coeliac disease).
10. Proliferative retinopathy.
11. Renal disease not associated with Type 1 Diabetes.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 443 (Actual)
Dates: Start 2009-01; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Albumin creatinine ratio | 2-4 years treatment duration
  The area under the curve over time of log ACR per year, with standardisation for gender, age and duration of disease

SECONDARY OUTCOMES:
Changes in CVD risk markers | 2-4 yrs treatment duration
  Changes in measures of:
  1. cIMT, FMD, EndoPAT and PWV between baseline and the end of intervention period;
  2. arterial BP, lipids and other lipoproteins, CVD risk markers (hsCRP and ADMA), assessed every 6 months during the intervention period.
Changes in glomerular filtration rate (GFR) | 2-4 years treatment duration
  Changes in measures of GFR (plasma SDMA, creatinine adn cystatin C levels) assessed every 6 months during intervention period.
Retinopathy | 2-4 years treatment duration
  Changes in retinopathy scores and retinal microvascular structure (arteriolar or venular dilation, vascular fractile dimension, branching and tortuosity) assessed annually
Quality of Life and Health Economics | 2-4 years treatment duration
  Changes in quality of life measures and resource usage

CONTACTS AND LOCATIONS:
Overall Officials: David B Dunger, Professor, Principal Investigator — University of Cambridge
Locations (2):
- University of Western Australia, Perth, Australia
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Amin R, Widmer B, Prevost AT, Schwarze P, Cooper J, Edge J, Marcovecchio L, Neil A, Dalton RN, Dunger DB. Risk of microalbuminuria and progression to macroalbuminuria in a cohort with childhood onset type 1 diabetes: prospective observational study. BMJ. 2008 Mar 29;336(7646):697-701. doi: 10.1136/bmj.39478.378241.BE. Epub 2008 Mar 18. PMID 18349042
- [Background] Dunger DB, Schwarze CP, Cooper JD, Widmer B, Neil HA, Shield J, Edge JA, Jones TW, Daneman D, Dalton RN. Can we identify adolescents at high risk for nephropathy before the development of microalbuminuria? Diabet Med. 2007 Feb;24(2):131-6. doi: 10.1111/j.1464-5491.2006.02047.x. PMID 17257274
- [Background] Adolescent type 1 Diabetes cardio-renal Intervention Trial Research Group. Adolescent type 1 Diabetes Cardio-renal Intervention Trial (AdDIT). BMC Pediatr. 2009 Dec 17;9:79. doi: 10.1186/1471-2431-9-79. PMID 20017932
- [Result] Cherney DZ, Scholey JW, Daneman D, Dunger DB, Dalton RN, Moineddin R, Mahmud FH, Dekker R, Elia Y, Sochett E, Reich HN. Urinary markers of renal inflammation in adolescents with Type 1 diabetes mellitus and normoalbuminuria. Diabet Med. 2012 Oct;29(10):1297-302. doi: 10.1111/j.1464-5491.2012.03651.x. PMID 22416821
- [Derived] Mahmud FH, Clarke ABM, Elia Y, Curtis J, Benitez-Aguirre P, Cameron FJ, Chiesa ST, Clarson C, Couper JJ, Craig ME, Dalton RN, Daneman D, Davis EA, Deanfield JE, Donaghue KC, Jones TW, Marshall SM, Neil A, Marcovecchio ML. Socioeconomic representativeness of Australian, Canadian and British cohorts from the paediatric diabetes AdDIT study: comparisons to regional and national data. BMC Med. 2023 Dec 20;21(1):506. doi: 10.1186/s12916-023-03222-w. PMID 38124088
- [Derived] Chiesa ST, Marcovecchio ML, Benitez-Aguirre P, Cameron FJ, Craig ME, Couper JJ, Davis EA, Dalton RN, Daneman D, Donaghue KC, Jones TW, Mahmud FH, Marshall SM, Neil HAW, Dunger DB, Deanfield JE; Adolescent Type 1 Diabetes Cardio-Renal Intervention Trial (AdDIT) Study Group. Vascular Effects of ACE (Angiotensin-Converting Enzyme) Inhibitors and Statins in Adolescents With Type 1 Diabetes. Hypertension. 2020 Dec;76(6):1734-1743. doi: 10.1161/HYPERTENSIONAHA.120.15721. Epub 2020 Oct 26. PMID 33100044
- [Derived] Niechcial E, Acerini CL, Chiesa ST, Stevens T, Dalton RN, Daneman D, Deanfield JE, Jones TW, Mahmud FH, Marshall SM, Neil HAW, Dunger DB, Marcovecchio ML; Adolescent Type 1 Diabetes Cardio-Renal Intervention Trial (AdDIT) Study Group; Adolescent Type 1 Diabetes Cardio-renal Intervention Trial AdDIT Study Group. Medication Adherence During Adjunct Therapy With Statins and ACE Inhibitors in Adolescents With Type 1 Diabetes. Diabetes Care. 2020 May;43(5):1070-1076. doi: 10.2337/dc19-0884. Epub 2020 Feb 27. PMID 32108022
- [Derived] Marcovecchio ML, Chiesa ST, Bond S, Daneman D, Dawson S, Donaghue KC, Jones TW, Mahmud FH, Marshall SM, Neil HAW, Dalton RN, Deanfield J, Dunger DB; AdDIT Study Group. ACE Inhibitors and Statins in Adolescents with Type 1 Diabetes. N Engl J Med. 2017 Nov 2;377(18):1733-1745. doi: 10.1056/NEJMoa1703518. PMID 29091568
- [Derived] Har RL, Reich HN, Scholey JW, Daneman D, Dunger DB, Moineddin R, Dalton RN, Motran L, Elia Y, Deda L, Ostrovsky M, Sochett EB, Mahmud FH, Cherney DZ. The urinary cytokine/chemokine signature of renal hyperfiltration in adolescents with type 1 diabetes. PLoS One. 2014 Nov 13;9(11):e111131. doi: 10.1371/journal.pone.0111131. eCollection 2014. PMID 25392936